CLINICAL TRIAL: NCT01885078
Title: A Phase 3, Multicenter Study to Evaluate the Long-Term Safety and Efficacy of Baricitinib in Patients With Rheumatoid Arthritis
Brief Title: An Extension Study in Participants With Moderate to Severe Rheumatoid Arthritis
Acronym: RA-BEYOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14060; I4V-MC-JADY (Other: Eli Lilly and Company); 2012-003686-17 (EudraCT Number)
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 4 milligram (mg) Baricitinib (Experimental): 4 mg Baricitinib administered orally once daily.
  Participants received baricitinib doses according to the dose received at the completion of the originating study. Participants may continue to receive the background non-investigational, open-label conventional disease-modifying antirheumatic drugs (cDMARD), nonsteroidal anti-inflammatory drug (NSAID), corticosteroid, and other analgesic therapies they were receiving at completion of the originating study.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 2 mg Baricitinib (Experimental): 2 mg Baricitinib administered orally once daily.
  Participants received baricitinib doses according to the dose received at the completion of the originating study. Participants may continue to receive the background non-investigational, open-label cDMARD, NSAID, corticosteroid, and other analgesic therapies they were receiving at completion of the originating study.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 2 mg Baricitinib Step-down (Experimental): 2 mg Baricitinib administered orally once daily in the 96-week Step-down period.
  Participants may continue to receive the background non-investigational, open-label cDMARD, NSAID, corticosteroid, and other analgesic therapies they were receiving at completion of the originating study.
  Interventions: Drug: Baricitinib
- 4 mg Baricitinib Step-down (Experimental): 4 mg Baricitinib administered orally once daily in the 96-week Step-down period.
  Participants may continue to receive the background non-investigational, open-label cDMARD, NSAID, corticosteroid, and other analgesic therapies they were receiving at completion of the originating study.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY 3009104; INCB 028050
Drug: Placebo — Administered orally
  Arms: 2 mg Baricitinib; 4 milligram (mg) Baricitinib

SUMMARY:
The purpose of this study is to investigate the long-term safety and any side effects of baricitinib in participants who have completed a previous baricitinib rheumatoid arthritis study.

The study provides 7 years of additional treatment with baricitinib.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the final active treatment in study JADV (NCT01710358), JADZ (NCT01711359), JADX (NCT01721057), JADW (NCT01721044), JADA (NCT01185353) or JAGS (NCT02265705)

Exclusion Criteria:

* Have significant uncontrolled cerebro-cardiovascular (eg, myocardial infarction [MI], unstable angina, unstable arterial hypertension, severe heart failure, or cerebrovascular accident), respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neuropsychiatric disorders, or abnormal laboratory values that developed during a previous baricitinib study that, in the opinion of the investigator, pose an unacceptable risk to the participant if investigational product continues to be administered
* Have a known hypersensitivity to baricitinib or any component of this investigational product
* Had investigational product permanently discontinued at any time during a previous baricitinib study
* Had temporary investigational product interruption at the final study visit of a previous baricitinib study and, in the opinion of the investigator, this poses an unacceptable risk for participation in the study
* Have any other condition that, in the opinion of the investigator, renders the participant unable to understand the nature, scope, and possible consequences of the study or precludes the participant from following and completing the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2877 (Actual)
Dates: Start 2013-06-27 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (408):
- United States (67):
  - Arizona Arthritis & Rheumatology Research, PLLC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Associates, P. C., Mesa, Arizona
  - Sun Valley Arthritis Center, LTD, Peoria, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Valley Endocrine, Fresno, Fresno, California
  - Allergy and Rheumatology Medical Clinic Inc, La Jolla, California
  - Desert Medical Advances, Palm Desert, California
  - Stanford University Hospital, Palo Alto, California
  - Pacific Arthritis Center, Santa Maria, California
  - Inland Rheumatology & Osteoporosis Medical Group, Upland, California
  - Boulder Medical Center, Boulder, Colorado
  - Denver Arthritis Clinic - Lowry, Denver, Colorado
  - New England Research Associates, Bridgeport, Connecticut
  - Clinical Research Center of CT/NY, Danbury, Connecticut
  - Delaware Arthritis, Lewes, Delaware
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Medallion Clinical Research Institute, Naples, Florida
  - Sun Coast Clinical Research, Inc, New Port Richey, Florida
  - Omega Research Consultants, Orlando, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Arthritis Research of Florida, Palm Harbor, Florida
  - West Broward Rheumatology Associates, Inc, Tamarac, Florida
  - AdventHealth Medical Group, Tampa, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Intermountain Research Center, Boise, Idaho
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Diagnostic Rheumatology and Research, Indianapolis, Indiana
  - Goldpoint Clinical Research LLC, Indianapolis, Indiana
  - Klein and Associates MD, PA, Cumberland, Maryland
  - West Michigan Rheumatology, Grand Rapids, Michigan
  - Borgess Rheumatology, Kalamazoo, Michigan
  - Advanced Rheumatology, PC, Lansing, Michigan
  - Office: Dr. Fiechtner, Justus, Lansing, Michigan
  - Arthritis and Osteporosis Treatment and Research Center, Flowood, Mississippi
  - University of Missouri, Columbia, Missouri
  - Clayton Medical Research, St Louis, Missouri
  - Arthritis Consultants, Inc., St Louis, Missouri
  - Dr. George Timothy Kelly, Las Vegas, Nevada
  - (AOA) Arthritis & Osteoporosis Associates, Freehold, New Jersey
  - Ocean Rheumatology, PA, Toms River, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - The Center for Rheumatology, Albany, New York
  - Drug Trials of America, Hartsdale, New York
  - Allergy Asthma Immunology of Rochester, AAIR Research Ctr, Rochester, New York
  - Asheville Rheumatology & Osteoporosis Research Assoc, PA, Asheville, North Carolina
  - Arthritis and Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Healthcare Research Consultant, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Arthritis Group, Philadelphia, Pennsylvania
  - Clinical Research Center of Reading,LLC, Wyomissing, Pennsylvania
  - Carolina Rheumatology and Neurology Associates, Myrtle Beach, South Carolina
  - Pioneer Research Solutions, Cypress, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Accurate Clinical Research, League City, Texas
  - Arthritis & Osteoporosis Associates LLP, Lubbock, Texas
  - Accurate Clinical Research, Webster, Texas
  - Center for Arthritis and Rheumatic Diseases, PC, Chesapeake, Virginia
  - Western Washington Arthritis Clinic, Bothell, Washington
  - Kadlec Clinic Rheumatology, Kennewick, Washington
  - The Vancouver Clinic, Vancouver, Washington
  - Rheumatology and Immunotherapy Center, Franklin, Wisconsin
- Argentina (27):
  - Hospital Italiano Regional del Sur, Bahía Blanca, Buenos Aires
  - Atencion Integral en Reumatología, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - CER Instituto Medico, Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Instituto Medico de Alta Complejidad San Isidro, San Isidro, Buenos Aires
  - CENIT Centro de Neurociencias, Investigación y Tratamiento, CABA, Ciudad Autonoma Buenos Aires
  - Instituto Centenario, CABA, Ciudad Autonoma de Buenos Aire
  - Centro de Enfermedades del Higado y Aparato Digestivo, Rosario, Santa Fe Province
  - Instituto CAICI SRL, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia, SAN M. de Tucuman, Tucumán Province
  - CIR Centro de Investigacions Reumatologicas, San Miguel de Tucumán, Tucumán Province
  - Consultorios Asociados de Endocrinologia, Ciudad Autonoma Buenos Aires
  - Organizacion Medica de Investigacion - OMI, Ciudad Autonoma de Buenos Aire
  - Centro De Osteopatias - Comlit, Ciudad Autonoma de Buenos Aire
  - Hospital Ramos Mejia, Ciudad Autonoma de Buenos Aire
  - Centro de Medicina Familiar Mindout Research, Ciudad Autonoma de Buenos Aire
  - Consultorios Reumatologicos Pampa, Ciudad Autonoma de Buenos Aire
  - CCBR Buenos Aires, Ciudad Autonoma de Buenos Aire
  - CEMIC Saavedra, Ciudad Autonoma de Buenos Aire
  - CENUDIAB, Ciudad Autonoma de Buenos Aire
  - Instituto Medico Strusberg, Córdoba
  - Hospital Italiano de Cordoba, Córdoba
  - Cent Priva Especiali Médicas Ambulatorias Inve Clin CEMAIC, Córdoba
  - Hospital Privado Centro Medico de Cordoba SA, Córdoba
  - Centro Polivalente de Asistencia e Inv. Clinica CER-San Juan, San Juan
- Australia (6):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Combined Rheumatology Practice (CRP), Kogarah, New South Wales
  - Coast Joint Care, Maroochydore, Queensland
  - Emeritus Research, Camberwell, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
- Austria (2):
  - Universitätsklinikum Graz, Graz, Styria
  - Rheuma Zentrum Favoriten GmbH, Vienna
- Belgium (5):
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - ZNA Jan Palfijn, Merksem, Flanders
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Reuma Clinic, Locatie Jaarbeurslaan, Genk
  - CHU Ambroise Pare, Mons
- Brazil (3):
  - CPCLIN, São Paulo, São Paulo
  - Associacao de Assistencia a Crianca Deficiente (AACD), São Paulo, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo, São Paulo
- Canada (12):
  - Rheumatology Research Associates Group, Edmonton, Alberta
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - Manitoba Clinic Medical Corporation, Winnipeg, Manitoba
  - KW Musculoskeletal Research Inc, Kitchener, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Peninsula Arthritis Centre, Inc., Saint Catherines, Ontario
  - UHN-Toronto Western Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Center de Recherche St Louis, Québec, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
  - Saskatoon Osteoporosis Centre, Saskatoon, Saskatchewan
- China (18):
  - Afflilated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliate Hospital of AnHui Medical University, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - 1st Hospital affiliated to Medical College of Shantou Univer, Shantou, Guangzhou
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - ZhuZhou Central Hospital, Zhuzhou, Hunan
  - YanCheng First People's Hospital, Yancheng, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Ningbo First Hospital, Ningbo, Zhejiang
  - China-Japan Friendship Hospital, Beijing
  - Shanghai Guanghua Hospital, Shanghai
- Croatia (3):
  - KBC Osijek, Osijek
  - Klinicka bolnica Sveti Duh, Zagreb
  - Poliklinika K-centar, Zagreb
- Czechia (9):
  - Revmatologicky ustav, Prague, Praha, Hlavní Mešto
  - Revmaclinic, s.r.o, Brno
  - Revmatologicka ambulance, Bruntál
  - ELIMATES BRNO s.r.o. Revmatologicka ambulance, Hustopeče
  - Vesalion s.r.o., Ostrava
  - Artroscan, s.r.o., Ostrava
  - ARTHROHELP s.r.o., Pardubice
  - Medical Plus, Uherské Hradiště
  - PV Medical Services s.r.o., Zlín
- Denmark (3):
  - Frederiksberg Hospital, Frederiksberg, Capital Region
  - Copenhagen University Hospital, Glostrup Municipality, Capital Region
  - Odense Universitetshospital, Odense C, Syd
- France (11):
  - CHRU de Limoges Hopital Dupuytren, Limoges, Haute-Vienne
  - Centre Hospitalier Jean Rougier, Cahors
  - Hôpital Trousseau, CHRU de Tours, Chambray-lès-Tours
  - Hôpital Arnaud de Villeneuve - CHU Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes
  - Nouvel Hôpital Orléans La Source, Orléans
  - Hopital de la Pitie Salpetriere, Paris
  - Hopital Cochin, Paris
  - CHU la Miletrie, Poitiers
  - CHU Rennes/Hopital Sud, Rennes
  - Hopital Bel Air, Thionville
- Germany (9):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Internistisch-rheumatologische Praxisgemeinschaft Bayreuth, Bayreuth, Bavaria
  - Klinikum der Universität München, München, Bavaria
  - Universitätsklinikum Würzburg A. ö. R., Würzburg, Bavaria
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Städtisches Klinikum Dresden-Friedrichstadt, Dresden, Saxony
  - Immunologisches Zentrum Vogelsang-Gommern GmbH, Gommern, Saxony-Anhalt
  - Charité Campus Virchow-Klinikum, Berlin
  - Schön Klinik Hamburg Eilbek, Hamburg
- Greece (4):
  - Hippokration Hospital of Athens, Athens, Attica
  - General Hospital of Attica KAT, Kifissia, Attica
  - University General Hospital of Heraklion, Heraklion, Crete
  - University General Hospital of Larissa, Larissa
- Hungary (7):
  - Dr. Rethy Pal Korhaz es Rendelointezet, Békéscsaba, Bekes County
  - Kiskunhalasi Semmelweis Korhaz, Kiskunhalas, Bács-Kiskun county
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár, Fejér
  - Revita Clinic, Budapest, Pest County
  - Szabolcs-Szatmar-Bereg M-i Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Orszagos Reumatologiai es Fizioterapias Intezet, Budapest
  - Csolnoky Ferenc Korhaz, Veszprém
- India (16):
  - Sumana Hospital, Hyderabad, Andhra Pradesh
  - Shalby Hospital, Ahmedabad, Gujarat
  - Medanta-The Medicity, Gurgaon, Haryana
  - Manipal Centre for Clinical Research (MCCR), Attavar, Mangalore, Karnataka
  - St. John Medical College & Hospital, Bangalore, Karnataka
  - M S Ramaiah Medical College Hospital, Bangalore, Karnataka
  - KLES Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - Kokilaben Dhirubhai Ambani Hospital &Medical Research Inst., Mumbai, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospital, New Delhi, National Capital Territory of Delhi
  - Shri Nidan Hospital & Hope Fertility Centre, Jaipur, Rajasthan
  - Care Hospital, Hyderabad, Telangana
  - Krishna Institute of Medical Sciences Ltd., Secunderabad, Telangana
  - CSM Medical University, Lucknow, Uttar Pradesh
  - IPGMER and SSKM Hospital, Kolkata, West Bengal
  - Apollo Gleneagles Hospitals Kolkata, Kolkata, West Bengal
- Israel (9):
  - Barzilai Medical Center, Ashkelon, Southern District
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin
  - Carmel Hospital, Haifa, Ḥeifā
- Italy (6):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Luigi Sacco, Milan
  - Stabilimento Ospedaliero Santa Chiara, Pisa
  - Polic.Umberto I -Univ. La Sapienza, Roma
  - Ospedale San Giovanni Bosco, Torino
  - Ospedale Policlinico Giambattista Rossi, Borgo Roma, Verona
- Japan (74):
  - Chubu-Rosai Hospital, Nagoya, Aichi-ken
  - Nagoya Medical Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Chiba-East-Hospital, Chuo-ku, Chiba
  - Matsudo City Hospital, Matsudo, Chiba
  - Chibaken Saiseikai Narashino Hospital, Narashino, Chiba
  - Shimoshizu National Hospital, Yotsukaidō, Chiba
  - PS Clinic, Hakata-ku, Fukuoka
  - Aso Iizuka Hospital, Iizuka, Fukuoka
  - University of Occupational and Enviromental Health, Kitakyushu, Fukuoka
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - Katayama Clinic, Asahikawa, Hokkaido
  - Sagawa Akira Rheumatology Clinic, Sapporo, Hokkaido
  - NTT East Japan Sapporo Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hokkaido Medical Center for Rheumatic Diseases, Sapporo, Hokkaido
  - Matsubara Mayflower Hospital, Katō, Hyōgo
  - Takarazuka City Hospital, Takarazuka, Hyōgo
  - Oasis Clinic, Hitachi, Ibaragi
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Yoshida Orthopaedic and Rheumatic Clinic, Morioka, Iwate
  - Komagamine Orthopedic and Rheumatology Clinic, Morioka, Iwate
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Yoshitama Clinic Rheumatology & Internal Medicine, Kirishima, Kagoshima-ken
  - Tokai University Hospital, Isehara, Kanagawa
  - St Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Yokohama Rosai Hospital, Yokohama, Kanagawa
  - Tsuzuki Azuma Clinic: Primary care and Rheumatology, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Yokohama Minami Kyosai Hospital, Yokohama, Kanagawa
  - Kumamoto Saishun Medical Center, Kōshi, Kumamoto
  - Yokkaichi Hazu Medical Center, Yokkaichi, Mie-ken
  - National Nagasaki Medical Center, Ōmura, Nagasaki
  - Sasebo Chuo Hospital, Sasebo, Nagasaki
  - Nagaoka Red Cross Hospital, Nagaoka, Niigata
  - Niigata Rheumatic Center, Shibata, Niigata
  - Osafune Clinic, Setouchi, Okayama-ken
  - Tomishiro Central Hospital, Tomigusuku, Okinawa
  - NHO Ureshino Medical Center, Ureshino, Saga-ken
  - Saitama Medical Center, Kawagoe, Saitama
  - Kaneko Clinic, Kawaguchi, Saitama
  - Azuma Rheumatology Clinic, Sayama, Saitama
  - Hirose Clinic, Tokorozawa, Saitama
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Women's Medical University East Medical Center, Arakawa-ku, Tokyo
  - St. Lukes International Hospital, Chuo-Ku, Tokyo
  - Fujimori Clinic, Hachiōji, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - National Tokyo Medical Center, Meguro-Ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Takaoka Rheumatic Orthopedic CL, Takaoka, Toyama
  - Miyasato Clinic, Shūnan, Yamaguchi
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kondo Clinic for Rheumatism and Orthopaedics, Fukuoka
  - Medical Co. LTA Fukuoka Mirai Hospital, Fukuoka
  - Shono Rheumatism Clinic, Fukuoka
  - Hiroshima Rheumatology Clinic, Hiroshima
  - Hiroshima Clinic, Hiroshima
  - Kagoshima Red Cross Hospital, Kagoshima
  - Kumamoto Rheumatology Clinic, Kumamoto
  - Kumamoto Orthopedic Hospital, Kumamoto
  - Kumamoto Shinto General hospital, Kumamoto
  - Nagano Red Cross Hospital, Nagano
  - Nagasaki Medical Hospital of Rheumatology, Nagasaki
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Okayama Saiseikai General Hospital Outpatient Center, Okayama
  - Okayama University Hospital, Okayama
  - Japanese Red Cross Okayama Hospital, Okayama
  - Yokota Clinic for Rheumatology, Osaka
  - Oribe Clinic Rheumatism and Medicine, Ōita
  - Shizuoka Rheumatism orthopedic Rehabilitation Hospital, Shizuoka
  - JA-Shizuoka Shizuoka-Kosei General Hospital, Shizuoka
- Latvia (3):
  - Rheumatology Practice in Jaunliepaja Primary Health Care Cen, Liepāja
  - Pauls Stradins Kliniska Universitates Slimnica, Riga
  - Dr. Sarmite Saleniece, Valmiera
- Lithuania (3):
  - Dr. Kildos Klinika, Kaunas
  - Klaipedos Universitetine Ligonine, Klaipėda
  - Respublikine Siauliu Ligonine, Šiauliai
- Mexico (16):
  - Ctro Inv en Artritis y Osteoporosis SC, Mexicali, Estado de Baja California
  - Centro de Investigacion del Noroeste, Tijuana, Estado de Baja California
  - Centro Integral en Reumatologia SA de CV, Guadalajara, Jalisco
  - Unidad de Investigacion en Enfermedades Cronico Degenerative, Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara, Jalisco
  - Private Service, Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Basica y Clinica, S.C., Guadalajara, Jalisco
  - Mexico Centre for Clinical Research SA de CV, Mexico City, Mexico City
  - RM Pharma Specialists S.A. de C.V., Mexico City, Mexico City
  - Hospital de Jesus I.A.P., Mexico City, Mexico City
  - Comite Mexicano para la Prevencion de la Osteoporosis A.C., Mexico City, Mexico City
  - Mentrials S.A. de C.V, Mexico City, Mexico City
  - Hospital Universitario de Monterrey, Monterrey, Nuevo León
  - Centro Medico de las Americas, Mérida, Yucatán
  - Medical Care and Research, S.A. de C.V., Mérida, Yucatán
  - Centro de Alta Especialidad Reumatologia e Inv Potosi, S.C., San Luis Potosí City
- Ziekenhuisgroep Twente, Almelo, Almelo, Netherlands
- Poland (8):
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Klinika Reumatologii i Ukladowych Chorob Tkanki Lacznej, Bydgoszcz
  - Ambulatorium Barbara Bazela, Elblag
  - Centrum Medyczne Pratia Katowice, Katowice
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - NZOZ Lecznica MAK-MED s.c., Nadarzyn
  - REUMATIKA - Centrum Reumatologii, Warsaw
  - Centrum Medyczne AMED, Warsaw
- Portugal (5):
  - Hospital Garcia da Orta, Almada
  - Instituto Portugues de Reumatologia, Lisbon
  - Hospital do Conde de Bertiandos, Ponte de Lima
  - Hospital Geral de Santo Antonio, Porto
  - Hospital de Sao Joao E.P.E., Porto
- Puerto Rico (5):
  - Ramon L. Ortega Colon, Carolina, PR
  - Ponce School of Medicine CAIMED Center, Ponce, PR
  - Latin Clinical Trial Center, San Juan, PR
  - Mindful Medical Research, San Juan, PR
  - Barbara Diaz Hernandez, San Juan, PR
- Romania (6):
  - Spital Clinic Judetean de Urgenta Tg.Mures, Tg.Mures, Mureș County
  - SC DUO Medical S.R.L Rheumatology, Bucharest
  - Spitalul Clinic Sf Maria Bucuresti, Bucharest
  - Spitalul Clinic "Dr. Ioan Cantacuzino", Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf.Apostol Andrei Constanta, Constanța
  - Spitalul Clinic de Recuperare Iasi, Iași
- Russia (10):
  - Gbuz Lokb, Saint-Petersburg, Leningradskaya Oblast'
  - GUZ UOKB, Ulyanovsk, Ulyanovsk Oblast
  - Family Clinic No 4, Korolyov
  - V.A. Nasonova Research Institute of Rheumatology, Moscow
  - City Clinical Hospital 1 named after N.I. Pirogov, Moscow
  - First Moscow State Medical University, Moscow
  - Ryazan Regional Clinincal Cardiology Dispensary, Ryazan
  - Clinical Rheumatology Hospital # 25, Saint Petersburg
  - Saratov Regional Clinical Hospital, Saratov
  - Clinical Emergency Hospital N.V.Solovyov, Yaroslavl
- Slovakia (5):
  - Nestatna reumatologicka ambulancia, Bratislava
  - ROMJAN s.r.o., Bratislava
  - Reumacentrum s.r.o., Partizánske
  - REUMED s.r.o., Spišská Nová Ves
  - LERAM s.r.o., Topoľčany
- Bolnisnica Dr. P. Drzaja UKCLJ, Ljubljana, Slovenia
- South Africa (6):
  - Netcare Greenacres Hospital, Port Elizabeth, Eastern Cape
  - Saint Augustine's Hospital, Durban, KZ-Natal
  - Precise Clinical Solutions (Pty) Ltd, Durban, KZ-Natal
  - Arthritis Clinical Trial Centre, Cape Town, Western Cape
  - Somerset West Trial Centre, Somerset West, Western Cape
  - Winelands Medical Research Centre, Stellenbosch, Western Cape
- South Korea (16):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Kyung Pook National University Hospital, Daegu, Korea
  - Daegu Catholic University Medical Center, Daegu, Korea
  - Chungnam National University Hospital, Daejeon, Korea
  - Chonnam National University Hospital, Gwangju, Korea
  - Gachon University Gil Medical Center, Incheon, Korea
  - Inha University Hospital, Incheon, Korea
  - Kyung Hee University Hospital, Seoul, Korea
  - Seoul National University Hospital, Seoul, Korea
  - Hanyang University Medical Center, Seoul, Korea
  - Kyunghee University Hospital at Gangdong, Seoul, Korea
  - Asan Medical Center, Seoul, Korea
  - Seoul St. Mary's Hospital, Seoul, Korea
  - Seoul Municipal Boramae Hospital, Seoul, Korea
  - Catholic University of Korea Yeouido St. Mary's Hospital, Seoul, Korea
  - Konkuk University Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (10):
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital Quiron Infanta Luisa, Seville, Andalusia
  - Corporacion Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques De Valdecilla, Santander, Cantabria
  - Hospital Universitario Getafe, Getafe, Madrid
  - Hospital De Basurto, Bilbao, Vizcaya
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario La Fe de Valencia, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Gothenburg
  - Reumatologiska Kliniken Skånes universitetssjukhus Malmö, Malmo
- Switzerland (3):
  - CHUV Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - HFR Fribourg - Hôpital Cantonal, Fribourg
  - Universitätsspital Zürich, Zurich
- Taiwan (9):
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - Tri-Service General Hospital, Neihu Taipei
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chi-Mei Medical Center, Yongkang District
- Trakya University, Edirne, Turkey (Türkiye)
- United Kingdom (7):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire
  - Southampton General Hospital, Southampton, Hants
  - Whipps Cross University Hospital, London, Surrey
  - Guy's Hospital, London, Surrey
  - Northumbria Healthcare NHS Foundation Trust, Newcastle upon Tyne, Tyneside
  - St Lukes Hospital, Bradford, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Caporali R, Taylor PC, Aletaha D, Sanmarti R, Takeuchi T, Mo D, Haladyj E, Bello N, Zaremba-Pechmann L, Fang Y, Dougados M. Efficacy of baricitinib in patients with moderate-to-severe rheumatoid arthritis up to 6.5 years of treatment: results of a long-term study. Rheumatology (Oxford). 2024 Oct 1;63(10):2799-2809. doi: 10.1093/rheumatology/keae012. PMID 38258434
- [Derived] Taylor PC, Takeuchi T, Burmester GR, Durez P, Smolen JS, Deberdt W, Issa M, Terres JR, Bello N, Winthrop KL. Safety of baricitinib for the treatment of rheumatoid arthritis over a median of 4.6 and up to 9.3 years of treatment: final results from long-term extension study and integrated database. Ann Rheum Dis. 2022 Mar;81(3):335-343. doi: 10.1136/annrheumdis-2021-221276. Epub 2021 Oct 27. PMID 34706874
- [Derived] Wells AF, Jia B, Xie L, Valenzuela GJ, Keystone EC, Li Z, Quebe AK, Griffing K, Otawa S, Haraoui B. Efficacy of Long-Term Treatment with Once-Daily Baricitinib 2 mg in Patients with Active Rheumatoid Arthritis: Post Hoc Analysis of Two 24-Week, Phase III, Randomized, Controlled Studies and One Long-Term Extension Study. Rheumatol Ther. 2021 Jun;8(2):987-1001. doi: 10.1007/s40744-021-00317-9. Epub 2021 May 24. PMID 34028703
- [Derived] Fleischmann R, Takeuchi T, Schiff M, Schlichting D, Xie L, Issa M, Stoykov I, Lisse J, Martinez-Osuna P, Rooney T, Zerbini CAF. Efficacy and Safety of Long-Term Baricitinib With and Without Methotrexate for the Treatment of Rheumatoid Arthritis: Experience With Baricitinib Monotherapy Continuation or After Switching From Methotrexate Monotherapy or Baricitinib Plus Methotrexate. Arthritis Care Res (Hoboken). 2020 Aug;72(8):1112-1121. doi: 10.1002/acr.24007. PMID 31233281
- [Derived] Tanaka Y, Fautrel B, Keystone EC, Ortmann RA, Xie L, Zhu B, Issa M, Patel H, Gaich CL, de Bono S, Rooney TP, Taylor PC. Clinical outcomes in patients switched from adalimumab to baricitinib due to non-response and/or study design: phase III data in patients with rheumatoid arthritis. Ann Rheum Dis. 2019 Jul;78(7):890-898. doi: 10.1136/annrheumdis-2018-214529. Epub 2019 Apr 30. PMID 31040122
- [Derived] Winthrop KL, Bingham CO 3rd, Komocsar WJ, Bradley J, Issa M, Klar R, Kartman CE. Evaluation of pneumococcal and tetanus vaccine responses in patients with rheumatoid arthritis receiving baricitinib: results from a long-term extension trial substudy. Arthritis Res Ther. 2019 Apr 18;21(1):102. doi: 10.1186/s13075-019-1883-1. PMID 30999933
- [Derived] Smolen JS, Genovese MC, Takeuchi T, Hyslop DL, Macias WL, Rooney T, Chen L, Dickson CL, Riddle Camp J, Cardillo TE, Ishii T, Winthrop KL. Safety Profile of Baricitinib in Patients with Active Rheumatoid Arthritis with over 2 Years Median Time in Treatment. J Rheumatol. 2019 Jan;46(1):7-18. doi: 10.3899/jrheum.171361. Epub 2018 Sep 15. PMID 30219772
- [Derived] Tanaka Y, McInnes IB, Taylor PC, Byers NL, Chen L, de Bono S, Issa M, Macias WL, Rogai V, Rooney TP, Schlichting DE, Zuckerman SH, Emery P. Characterization and Changes of Lymphocyte Subsets in Baricitinib-Treated Patients With Rheumatoid Arthritis: An Integrated Analysis. Arthritis Rheumatol. 2018 Dec;70(12):1923-1932. doi: 10.1002/art.40680. Epub 2018 Oct 22. PMID 30058112
- [Derived] Taylor PC, Kremer JM, Emery P, Zuckerman SH, Ruotolo G, Zhong J, Chen L, Witt S, Saifan C, Kurzawa M, Otvos JD, Connelly MA, Macias WL, Schlichting DE, Rooney TP, de Bono S, McInnes IB. Lipid profile and effect of statin treatment in pooled phase II and phase III baricitinib studies. Ann Rheum Dis. 2018 Jul;77(7):988-995. doi: 10.1136/annrheumdis-2017-212461. Epub 2018 Feb 20. PMID 29463520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible to participate in the Step-down period if they achieved a sustained (at least 3 months in JADY) low disease activity (CDAI score ≤10; for participants originating in Studies JADV, JADX, JADW, and JAGS) or sustained remission (CDAI score ≤2.8; for participants originating in Study JADZ). Eligible participants were randomized to 4 mg or 2 mg baricitinib once daily to evaluate if treatment with 2 mg maintains the low disease activity achieved with 4 mg baricitinib.
Pre-assignment Details: Participants who completed an originating study:
  I4V-MC-JADZ (NCT01711359), I4V-MC-JADV (NCT017103580, I4V-MC-JADX (NCT01721057), I4V-MC-JADW (NCT01721044), I4V-MC-JADA (NCT01185353), or I4V-MC-JAGS (NCT02265705) were eligible for enrollment into study JADY.
Groups:
- JADZ 4 Milligram (mg) Baricitinib; JADV 4 mg Baricitinib; JADX 4 mg Baricitinib; JADW 4 mg Baricitinib; JAGS 4 mg Baricitinib; JADA 4 mg Baricitinib: 4 mg Baricitinib administered orally once daily.
- JADX 2 mg Baricitinib; JADW 2 mg Baricitinib: 2 mg Baricitinib administered orally once daily.
- 2 mg Baricitinib Step-down: 2 mg Baricitinib administered orally once daily in the 96-week Step-down period.
- 4 mg Baricitinib Step-down: 4 mg Baricitinib administered orally once daily in the 96-week Step-down period.
Period: Treatment Period
Arm/Group | JADZ 4 Milligram (mg) Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib | 2 mg Baricitinib Step-down | 4 mg Baricitinib Step-down
Started | 451 | 1091 | 180 | 403 | 117 | 331 | 221 | 83 | 0 | 0
Received at Least Once Dose of Study Drug | 451 | 1090 | 180 | 403 | 117 | 331 | 221 | 83 | 0 | 0
Completed | 19 | 64 | 49 | 120 | 27 | 81 | 0 | 55 | 0 | 0
Not Completed | 432 | 1027 | 131 | 283 | 90 | 250 | 221 | 28 | 0 | 0
Not completed — Adverse Event | 52 | 136 | 30 | 73 | 17 | 72 | 24 | 5 | 0 | 0
Not completed — Death | 13 | 33 | 5 | 9 | 2 | 10 | 3 | 2 | 0 | 0
Not completed — Lack of Efficacy | 12 | 33 | 10 | 23 | 24 | 58 | 9 | 5 | 0 | 0
Not completed — Lost to Follow-up | 16 | 19 | 7 | 9 | 2 | 8 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 19 | 21 | 5 | 12 | 9 | 24 | 4 | 3 | 0 | 0
Not completed — Protocol Violation | 3 | 5 | 0 | 3 | 1 | 6 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 245 | 648 | 49 | 90 | 20 | 38 | 162 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 72 | 132 | 25 | 63 | 15 | 34 | 17 | 10 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step-down Period
Arm/Group | JADZ 4 Milligram (mg) Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib | 2 mg Baricitinib Step-down | 4 mg Baricitinib Step-down
Started | 0 (Not all participants were eligible to enter the Step-Down Period.) | 0 (Not all participants were eligible to enter the Step-Down Period.) | 0 (Not all participants were eligible to enter the Step-Down Period.) | 0 (Not all participants were eligible to enter the Step-Down Period.) | 0 (Not all participants were eligible to enter the Step-Down Period.) | 0 (Not all participants were eligible to enter the Step-Down Period.) | 0 | 0 (Not all participants were eligible to enter the Step-Down Period.) | 592 (Eligible participants were offered the option of participating in the Step-Down Period.) | 594 (Eligible participants were offered the option of participating in the Step-Down Period.)
Complete Through Week 96 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 407 | 455
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 523 | 533
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 69 | 61
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 38
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 15
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- JADZ 4 mg Baricitinib; JADV 4 mg Baricitinib; JADX 4 mg Baricitinib; JADW 4 mg Baricitinib; JAGS 4 mg Baricitinib; JADA 4 mg Baricitinib: 4 mg Baricitinib administered orally once daily.
- Total: Total of all reporting groups
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib | Total
Number analyzed (Participants) | 451 | 1090 | 180 | 403 | 117 | 331 | 221 | 83 | 2876
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 386 | 881 | 150 | 335 | 86 | 253 | 199 | 68 | 2358
  >=65 years | 65 | 209 | 30 | 68 | 31 | 78 | 22 | 15 | 518
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 326 | 847 | 144 | 335 | 87 | 275 | 177 | 71 | 2262
  Male | 125 | 243 | 36 | 68 | 30 | 56 | 44 | 12 | 614
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 35 | 56 | 1 | 12 | 6 | 21 | 6 | 6 | 143
  Asian | 122 | 321 | 50 | 94 | 6 | 19 | 167 | 2 | 781
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 17 | 4 | 9 | 10 | 7 | 12 | 3 | 2 | 64
  White | 275 | 691 | 119 | 283 | 98 | 275 | 45 | 73 | 1859
  More than one race | 2 | 17 | 1 | 2 | 0 | 1 | 0 | 0 | 23
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68 | 64 | 39 | 103 | 52 | 136 | 0 | 26 | 488
  Czechia | 0 | 29 | 3 | 10 | 0 | 0 | 0 | 14 | 56
  Portugal | 3 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 11
  Russia | 35 | 70 | 10 | 7 | 0 | 0 | 0 | 0 | 122
  Greece | 0 | 2 | 0 | 0 | 2 | 4 | 0 | 0 | 8
  South Korea | 6 | 43 | 6 | 8 | 3 | 6 | 0 | 0 | 72
  Latvia | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Sweden | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Austria | 2 | 0 | 0 | 0 | 3 | 12 | 0 | 0 | 17
  Netherlands | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  China | 0 | 41 | 0 | 0 | 0 | 0 | 167 | 0 | 208
  Poland | 0 | 66 | 11 | 37 | 9 | 22 | 0 | 11 | 156
  Brazil | 16 | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 30
  Slovenia | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Slovakia | 0 | 17 | 3 | 7 | 0 | 0 | 0 | 0 | 27
  France | 0 | 16 | 0 | 0 | 6 | 14 | 0 | 0 | 36
  Lithuania | 0 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 21
  Croatia | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 6 | 9
  Argentina | 87 | 226 | 15 | 44 | 3 | 15 | 40 | 0 | 430
  Romania | 0 | 14 | 2 | 2 | 0 | 0 | 0 | 3 | 21
  Hungary | 0 | 30 | 8 | 11 | 0 | 0 | 0 | 11 | 60
  Japan | 82 | 215 | 4 | 13 | 3 | 11 | 0 | 0 | 328
  United Kingdom | 10 | 8 | 3 | 1 | 1 | 3 | 0 | 0 | 26
  Switzerland | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 7
  India | 28 | 0 | 16 | 27 | 0 | 0 | 0 | 0 | 71
  Spain | 0 | 28 | 9 | 24 | 6 | 19 | 0 | 0 | 86
  Canada | 13 | 8 | 8 | 13 | 3 | 2 | 0 | 0 | 47
  Turkey | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3
  Belgium | 20 | 7 | 3 | 8 | 0 | 3 | 0 | 0 | 41
  Taiwan | 0 | 12 | 23 | 46 | 0 | 0 | 0 | 0 | 81
  Denmark | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 5
  South Africa | 16 | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 56
  Italy | 12 | 0 | 3 | 6 | 3 | 3 | 0 | 0 | 27
  Mexico | 39 | 115 | 8 | 14 | 5 | 21 | 0 | 12 | 214
  Israel | 0 | 0 | 0 | 0 | 6 | 21 | 0 | 0 | 27
  Australia | 0 | 0 | 1 | 12 | 5 | 14 | 0 | 0 | 32
  Germany | 11 | 2 | 1 | 6 | 3 | 13 | 0 | 0 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events (AEs) or Serious AE
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (i.e., abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Non-serious AEs are reported at a threshold of 5%.
  An SAE is an AE from this study that results in any of the following: death, initial or prolonged inpatient hospitalization, a life-threatening experience, persistent or significant disability/incapacity, congenital anomaly/birth defect, considered significant by the investigator for any other reason
  A summary of serious adverse events (SAEs) and other non-serious adverse events (AEs), regardless of causality, were reported in the Reported Adverse Events module.
Time Frame: Baseline through 84 Months
Population: All enrolled participants who received at least one dose of study drug and did not discontinue the study for the reason 'Lost to Follow-up' at the first postbaseline visit in study JADY.
Measure: Number; unit: participants
Groups:
- 2 mg Baricitinib: 2 mg Baricitinib administered orally once daily.
- 4 mg Baricitinib: 4 mg Baricitinib administered orally once daily.
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | 2 mg Baricitinib Step-down | 4 mg Baricitinib Step-down
Number analyzed (Participants) | 297 | 2579 | 592 | 594
participants
  Adverse Events | 234 | 1532 | 270 | 315
  Serious Adverse Events | 112 | 517 | 164 | 178

2. Secondary Outcome: Percentage of Participants Maintaining an American College of Rheumatology (ACR) Response of ACR20
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis (RA). An ACR20 Responder is a participant who had ≥20% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessment of participant's physical function), pain due to RA, and hsCRP. Percentage of participants achieving ACR20 response = (number of ACR20 responders) / (number of participants analyzed) * 100
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
Percentage of Participants | 92.6 [89.7 to 94.7] | 88.4 [86.3 to 90.2] | 79.3 [72.6 to 84.7] | 79.5 [75.1 to 83.3] | 72.3 [62.9 to 80.1] | 70.8 [65.2 to 75.9] | 86.7 [81.4 to 90.6] | 75.6 [65.1 to 83.8]

3. Secondary Outcome: Percentage of Participants Maintaining an American College of Rheumatology (ACR) Response of ACR20
Description: as for outcome 2
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 78.3 [74.1 to 82.0] | 76.6 [73.9 to 79.1] | 71.6 [64.4 to 77.9] | 70.5 [65.6 to 74.9] | 57.4 [47.7 to 66.6] | 55.8 [49.9 to 61.6] | 73.8 [67.5 to 79.3] | 71.8 [61.0 to 80.6]

4. Secondary Outcome: Percentage of Participants Maintaining an American College of Rheumatology (ACR) Response of ACR20
Description: as for outcome 2
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 67.3 [62.7 to 71.6] | 65.6 [62.6 to 68.4] | 60.4 [52.8 to 67.4] | 56.0 [50.9 to 61.0] | 50.5 [40.9 to 60.0] | 43.1 [37.3 to 49.0] | 24.8 [19.4 to 31.0] | 60.3 [49.2 to 70.4]

5. Secondary Outcome: Percentage of Participants Maintaining an American College of Rheumatology (ACR) Response of ACR50
Description: ACR50 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis (RA). An ACR50 Responder is a participant who had ≥50% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥50% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessment of participant's physical function), pain due to RA, and hsCRP. Percentage of participants achieving ACR50 response = (number of ACR50 responders) / (number of participants analyzed) * 100
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 80.0 [75.9 to 83.5] | 67.7 [64.8 to 70.5] | 58.0 [50.5 to 65.2] | 58.2 [53.1 to 63.1] | 45.5 [36.2 to 55.2] | 43.8 [38.0 to 49.7] | 69.0 [62.5 to 74.9] | 43.6 [33.1 to 54.6]

6. Secondary Outcome: Percentage of Participants Maintaining an American College of Rheumatology (ACR) Response of ACR50
Description: as for outcome 5
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 67.8 [63.2 to 72.1] | 61.6 [58.6 to 64.5] | 49.7 [42.3 to 57.2] | 53.3 [48.2 to 58.3] | 43.6 [34.3 to 53.3] | 36.5 [31.0 to 42.3] | 59.0 [52.3 to 65.5] | 43.6 [33.1 to 54.6]

7. Secondary Outcome: Percentage of Participants Maintaining an American College of Rheumatology (ACR) Response of ACR50
Description: as for outcome 5
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 59.9 [55.1 to 64.5] | 52.7 [49.7 to 55.7] | 44.4 [37.1 to 51.9] | 43.2 [38.2 to 48.3] | 37.6 [28.8 to 47.4] | 32.1 [26.9 to 37.9] | 18.6 [13.9 to 24.4] | 37.2 [27.3 to 48.3]

8. Secondary Outcome: Percentage of Participants Maintaining an American College of Rheumatology (ACR) Response of ACR70
Description: ACR70 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis (RA). An ACR70 Responder is a participant who had ≥70% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥70% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessment of participant's physical function), pain due to RA, and hsCRP. Percentage of participants achieving ACR70 response = (number of ACR70 responders) / (number of participants analyzed) * 100
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 61.3 [56.6 to 65.9] | 45.7 [42.7 to 48.8] | 34.9 [28.1 to 42.4] | 35.8 [31.1 to 40.8] | 28.7 [20.8 to 38.2] | 25.9 [21.1 to 31.4] | 42.9 [36.4 to 49.6] | 26.9 [18.3 to 37.7]

9. Secondary Outcome: Percentage of Participants Maintaining an American College of Rheumatology (ACR) Response of ACR70
Description: as for outcome 8
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 54.4 [49.6 to 59.1] | 44.1 [41.1 to 47.1] | 35.5 [28.7 to 43.0] | 32.5 [27.9 to 37.5] | 24.8 [17.4 to 34.0] | 21.5 [17.1 to 26.8] | 35.2 [29.1 to 41.9] | 21.8 [14.1 to 32.2]

10. Secondary Outcome: Percentage of Participants Maintaining an American College of Rheumatology (ACR) Response of ACR70
Description: as for outcome 8
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 Milligram (mg) Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 48.2 [43.5 to 53.0] | 39.1 [36.1 to 42.1] | 28.4 [22.1 to 35.6] | 28.4 [24.0 to 33.2] | 23.8 [16.5 to 32.9] | 18.2 [14.1 to 23.2] | 12.9 [9.0 to 18.1] | 19.2 [12.0 to 29.3]

11. Secondary Outcome: Percentage of Participants Maintaining a Disease Activity Score (DAS28) High-Sensitivity C-Reactive Protein (hsCRP) ≤3.2
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count-28 (TJC28), swollen joint count-28 (SJC28), CRP (mg/L), and Patient's Global Assessment of Disease Activity using VAS (patient's global VAS). DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*patient's global VAS+0.96. Scores ranged from 1.0-9.4, where lower scores indicated less disease activity, low disease activity was DAS28-CRP ≤3.2 and remission was DAS28-CRP <2.6. A decrease in DAS28-CRP indicated an improvement in participant's condition.
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 81.9 [77.9 to 85.3] | 71.9 [69.0 to 74.5] | 66.3 [58.9 to 73.0] | 68.6 [63.7 to 73.1] | 50.5 [40.9 to 60.0] | 51.1 [45.2 to 57.0] | 72.4 [66.0 to 78.0] | 59.0 [47.9 to 69.2]

12. Secondary Outcome: Percentage of Participants Maintaining a Disease Activity Score (DAS28) High-Sensitivity C-Reactive Protein (hsCRP) ≤3.2
Description: as for outcome 11
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 71.8 [67.3 to 75.9] | 65.5 [62.5 to 68.3] | 59.2 [51.6 to 66.3] | 59.3 [54.2 to 64.2] | 47.5 [38.1 to 57.2] | 41.6 [35.9 to 47.5] | 61.0 [54.2 to 67.3] | 60.3 [49.2 to 70.4]

13. Secondary Outcome: Percentage of Participants Maintaining a Disease Activity Score (DAS28) High-Sensitivity C-Reactive Protein (hsCRP) ≤3.2
Description: as for outcome 11
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 61.1 [56.3 to 65.6] | 58.9 [55.9 to 61.9] | 46.7 [39.4 to 54.3] | 50.0 [44.9 to 55.1] | 44.6 [35.2 to 54.3] | 34.3 [28.9 to 40.1] | 21.0 [16.0 to 27.0] | 53.8 [42.9 to 64.5]

14. Secondary Outcome: Percentage of Participants Maintaining a Disease Activity Score (DAS28) High-Sensitivity C-Reactive Protein (hsCRP)<2.6
Description: as for outcome 11
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 Milligram (mg) Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 65.6 [61.0 to 70.0] | 52.3 [49.3 to 55.4] | 50.9 [43.4 to 58.3] | 46.2 [41.1 to 51.3] | 34.7 [26.1 to 44.3] | 32.8 [27.6 to 38.6] | 52.4 [45.6 to 59.0] | 44.9 [34.3 to 55.9]

15. Secondary Outcome: Percentage of Participants Maintaining a Disease Activity Score (DAS28) High-Sensitivity C-Reactive Protein (hsCRP)<2.6
Description: as for outcome 11
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 59.9 [55.1 to 64.5] | 51.0 [47.9 to 54.0] | 43.8 [36.5 to 51.3] | 43.2 [38.2 to 48.3] | 31.7 [23.4 to 41.3] | 26.3 [21.4 to 31.8] | 38.6 [32.2 to 45.3] | 35.9 [26.1 to 47.0]

16. Secondary Outcome: Percentage of Participants Maintaining a Disease Activity Score (DAS28) High-Sensitivity C-Reactive Protein (hsCRP)<2.6
Description: as for outcome 11
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 51.1 [46.3 to 55.8] | 44.0 [41.0 to 47.0] | 36.1 [29.2 to 43.6] | 37.7 [32.9 to 42.8] | 29.7 [21.7 to 39.2] | 26.6 [21.8 to 32.2] | 13.3 [9.4 to 18.6] | 43.6 [33.1 to 54.6]

17. Secondary Outcome: Percentage of Participants Maintaining a DAS28-Erythrocyte Sedimentation Rate (ESR) Score of ≤3.2
Description: DAS28 consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), ESR (millimeters per hour), and Patient's Global Assessment of Disease Activity. DAS28 was calculated using following formula: DAS28-ESR=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.70*natural log(ESR)+0.014*Patient's Global VAS. Total scores ranged from 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 61.8 [57.1 to 66.3] | 48.4 [45.3 to 51.4] | 46.2 [38.8 to 53.7] | 48.4 [43.3 to 53.5] | 31.7 [23.4 to 41.3] | 31.8 [26.5 to 37.5] | 41.0 [34.5 to 47.7] | 35.9 [26.1 to 47.0]

18. Secondary Outcome: Percentage of Participants Maintaining a DAS28-Erythrocyte Sedimentation Rate (ESR) Score of ≤3.2
Description: as for outcome 17
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 54.4 [49.6 to 59.1] | 46.1 [43.1 to 49.2] | 40.2 [33.1 to 47.8] | 41.0 [36.1 to 46.1] | 22.8 [15.7 to 31.9] | 23.7 [19.1 to 29.1] | 33.8 [27.8 to 40.4] | 37.2 [27.3 to 48.3]

19. Secondary Outcome: Percentage of Participants Maintaining a DAS28-Erythrocyte Sedimentation Rate (ESR) Score of ≤3.2
Description: as for outcome 17
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 48.7 [43.9 to 53.5] | 41.3 [38.3 to 44.3] | 36.1 [29.2 to 43.6] | 32.5 [27.9 to 37.5] | 23.8 [16.5 to 32.9] | 21.9 [17.4 to 27.2] | 11.4 [7.8 to 16.4] | 37.2 [27.3 to 48.3]

20. Secondary Outcome: Percentage of Participants Maintaining a DAS28-Erythrocyte Sedimentation Rate (ESR) Sore of <2.6
Description: as for outcome 17
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 36.8 [32.3 to 41.5] | 29.3 [26.6 to 32.2] | 24.3 [18.4 to 31.2] | 26.8 [22.5 to 31.5] | 20.8 [14.0 to 29.7] | 13.1 [9.6 to 17.7] | 25.2 [19.8 to 31.5] | 15.4 [9.0 to 25.0]

21. Secondary Outcome: Percentage of Participants Maintaining a DAS28-Erythrocyte Sedimentation Rate (ESR) Sore of <2.6
Description: as for outcome 17
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 38.9 [34.4 to 43.7] | 24.7 [22.1 to 27.4] | 24.3 [18.4 to 31.2] | 23.2 [19.2 to 27.8] | 15.8 [10.0 to 24.2] | 10.2 [7.2 to 14.4] | 19.5 [14.7 to 25.4] | 23.1 [15.1 to 33.6]

22. Secondary Outcome: Percentage of Participants Maintaining a DAS28-Erythrocyte Sedimentation Rate (ESR) Sore of <2.6
Description: as for outcome 17
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 31.3 [27.0 to 35.9] | 23.9 [21.4 to 26.6] | 22.5 [16.8 to 29.4] | 19.4 [15.7 to 23.8] | 11.9 [6.9 to 19.6] | 8.8 [6.0 to 12.7] | 7.1 [4.4 to 11.4] | 19.2 [12.0 to 29.3]

23. Secondary Outcome: Percentage of Participants Maintaining American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Boolean Remission Response
Description: Boolean-based definition of remission, all 4 criteria below must be met: tender joint count (TJC28 ) <=1, swollen joint count (SJC28) <=1, hsCRP <=1 milligram per deciliter (mg/dL), Patient Global Assessment of Disease Activity using visual analog scale (VAS) <=1 cm.
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 30.5 [26.3 to 35.1] | 20.8 [18.4 to 23.4] | 17.8 [12.7 to 24.2] | 17.8 [14.2 to 22.0] | 8.9 [4.8 to 16.1] | 9.5 [6.6 to 13.5] | 17.1 [12.6 to 22.8] | 12.8 [7.1 to 22.0]

24. Secondary Outcome: Percentage of Participants Maintaining American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Boolean Remission Response
Description: as for outcome 23
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 30.8 [26.6 to 35.4] | 20.3 [18.0 to 22.9] | 16.6 [11.7 to 22.9] | 15.0 [11.7 to 19.1] | 9.9 [5.5 to 17.3] | 8.0 [5.4 to 11.9] | 11.9 [8.2 to 17.0] | 15.4 [9.0 to 25.0]

25. Secondary Outcome: Percentage of Participants Maintaining American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Boolean Remission Response
Description: as for outcome 23
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 26.5 [22.5 to 30.9] | 17.7 [15.5 to 20.1] | 13.6 [9.2 to 19.6] | 14.2 [11.0 to 18.2] | 6.9 [3.4 to 13.6] | 7.3 [4.8 to 11.0] | 5.2 [2.9 to 9.1] | 15.4 [9.0 to 25.0]

26. Secondary Outcome: Change From Baseline of Originating Study in Modified Total Sharp Score (mTSS)
Description: X-rays of the hands/wrists and feet were scored for structural progression as measured using the mTSS. This methodology quantified the extent of bone erosions and joint space narrowing (JSN) for 44 and 42 joints, with higher scores representing greater damage. The mTSS at a time point is the sum of the erosion (range from 0 to 280) and JSN (range from 0 to 168) scores, for a maximum score of 448. Least Squares Mean (LSM) was calculated using a mixed model for repeated measures (MMRM) with treatment, visit, treatment-by-visit-interactions as fixed categorical effects and baseline and baseline-by-visit-interactions as fixed continuous effects.
Time Frame: Baseline, Year 1
Population: All enrolled participants who received at least one dose of study drug in JADY with available baseline x-ray (from originating study) and at least 1 postbaseline x-ray assessment (collected in JADY) and Year 1 data. Zero participants analyzed, no data collected in this study or originating study.
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Change From Baseline of Originating Study in Modified Total Sharp Score (mTSS)
Description: as for outcome 26
Time Frame: Baseline, Year 3
Population: All enrolled participants treated with at least one dose of study drug in JADY with available baseline x-ray (from originating study) and at least 1 postbaseline x-ray assessment (collected in JADY) and Year 3 data. JADW and JADA, zero participants analyzed due to no data collected in this study or originating study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 387 | 343 | 137 | 301 | 0 | 0 | 203 | 0
score on a scale | 1.30 [0.94 to 1.67] | 1.64 [1.38 to 1.90] | 1.13 [0.61 to 1.66] | 1.13 [0.78 to 1.48] |  |  | 1.20 [0.61 to 1.80] |

28. Secondary Outcome: Change From Baseline of Originating Study in Modified Total Sharp Score (mTSS)
Description: as for outcome 26
Time Frame: Baseline, Year 5
Population: All enrolled participants treated with at least one dose of study drug in JADY with available baseline x-ray (from originating study) and at least 1 postbaseline x-ray assessment (collected in JADY) and Year 5 data. JAGS, JADW and JADA, zero participants analyzed due to no data collected in this study or originating study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 349 | 870 | 127 | 276 | 0 | 0 | 0 | 0
score on a scale | 1.64 [1.18 to 2.09] | 2.18 [1.85 to 2.51] | 1.32 [0.69 to 1.96] | 1.58 [1.15 to 2.02] |  |  |  |

29. Secondary Outcome: Percentage of Participants With mTSS Change ≤0
Description: X-rays of the hands/wrists and feet were scored for structural progression as measured using the mTSS. This methodology quantified the extent of bone erosions and joint space narrowing (JSN) for 44 and 42 joints, with higher scores representing greater damage. The mTSS at a time point is the sum of the erosion (range from 0 to 280) and JSN (range from 0 to 168) scores, for a maximum score of 448, with higher scores representing greater damage.
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY. Year 1 data not available, zero participants analyzed due to no data collected in this study or originating study.
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Percentage of Participants With mTSS Change ≤0
Description: as for outcome 29
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY. JADW and JADA, zero participants analyzed due to no data collected in this study or originating study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 0 | 0 | 210 | 0
percentage of participants | 53.5 [48.7 to 58.2] | 53.0 [50.0 to 56.0] | 0.6 [0.1 to 3.3] | 0.8 [0.3 to 2.4] |  |  | 0 [0.0 to 1.8] |

31. Secondary Outcome: Percentage of Participants With mTSS Change ≤0
Description: as for outcome 29
Time Frame: Year 5 after entry into JADY
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 0 | 0 | 210 | 0
percentage of participants | 1.7 [0.8 to 3.4] | 0.6 [0.3 to 1.3] | 0 [0.0 to 2.2] | 0.5 [0.1 to 2.0] |  |  | 0 [0.0 to 1.8] |

32. Secondary Outcome: Change From Baseline of Originating Study in Joint Space Narrowing at Year 1
Description: X-rays of the hands/wrists and feet were assessed for joint space narrowing (JSN) and bone erosions. Assessment of JSN for each hand (15 joints per hand) and foot (6 joints per foot), including subluxation, is scored from 0 to 4, with 0 indicating no (normal) JSN and 4 indicating complete loss of joint space, bony ankylosis or luxation. JSN scores ranged from 0-168. A score of 0 would indicate no change and higher scores represent a worsening of joint space narrowing.
Time Frame: Baseline, Year 1
Population: All enrolled participants treated with at least one dose of study drug in JADY with available baseline (from originating study) and at least 1 postbaseline x-ray assessment (collected in JADY). Year 1 data not available, zero participants analyzed due to no data collected in this study or originating study.
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

33. Secondary Outcome: Change From Baseline of Originating Study in Joint Space Narrowing at Year 3
Description: as for outcome 32
Time Frame: Baseline, Year 3
Population: All enrolled participants treated with at least one dose of study drug in JADY with available baseline (from originating study) and at least 1 postbaseline x-ray assessment (collected in JADY). JADW and JADA, zero participants analyzed due to no data collected in this study or originating study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 387 | 943 | 137 | 301 | 0 | 0 | 203 | 0
score on a scale | 0.45 [0.26 to 0.63] | 0.72 [0.59 to 0.86] | 0.54 [0.25 to 0.83] | 0.44 [0.24 to 0.63] |  |  | 0.52 [0.23 to 0.82] |

34. Secondary Outcome: Change From Baseline of Originating Study in Joint Space Narrowing at Year 5
Description: as for outcome 32
Time Frame: Baseline, Year 5
Population: All enrolled participants treated with at least one dose of study drug in JADY with available baseline (from originating study) and at least 1 postbaseline x-ray assessment (collected in JADY). JAGS, JADW, and JADA, zero participants analyzed due to no data collected in this study or originating study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 349 | 870 | 127 | 276 | 0 | 0 | 0 | 0
score on a scale | 0.59 [0.36 to 0.83] | 1.00 [0.84 to 1.17] | 0.68 [0.34 to 1.02] | 0.60 [0.37 to 0.83] |  |  |  |

35. Secondary Outcome: Change From Baseline of Originating Study in Duration of Morning Stiffness
Description: Participants reported the duration of their morning joint stiffness (MJS) in hours and minutes. The participants were asked about their duration of morning joint stiffness on the day prior to the study visit to capture actual symptoms, since the participant may have had an atypical morning routine on the day of the study visit. If morning joint stiffness duration was longer than 12 hours (720 minutes), it was truncated to 720 minutes for statistical presentations and analyses. A decrease in duration of morning joint stiffness indicated an improvement in the participant's condition.
Time Frame: Baseline, Year 1
Population: All enrolled participants who received at least one dose of study drug in JADY and had evaluable morning stiffness data. Data not collected for JADX; zero participants analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 450 | 633 | 0 | 0 | 110 | 308 | 221 | 78
minutes | -102.72 (155.27) | -73.53 (144.22) |  |  | -75.07 (139.00) | -73.88 (149.55) | -68.74 (148.34) | -37.12 (61.34)

36. Secondary Outcome: Change From Baseline of Originating Study in Duration of Morning Stiffness
Description: as for outcome 35
Time Frame: Baseline, Year 3
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 387 | 556 | 0 | 0 | 81 | 222 | 192 | 69
minutes | -112.41 (159.78) | -77.78 (141.01) |  |  | -84.60 (127.85) | -67.79 (154.05) | -90.61 (147.70) | -47.13 (52.97)

37. Secondary Outcome: Change From Baseline of Originating Study in Duration of Morning Stiffness
Description: as for outcome 35
Time Frame: Baseline, Year 5
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | JADZ 4 Milligram (mg) Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 330 | 470 | 0 | 0 | 70 | 169 | 128 | 57
minutes | -111.45 (164.74) | -82.48 (137.23) |  |  | -88.37 (146.73) | -91.57 (163.88) | -92.75 (125.39) | -45.89 (60.43)

38. Secondary Outcome: Change From Baseline of Originating Study in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Health State Scores
Description: The European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) is a standardized measure of health status of the participant. The first component is a descriptive system of the respondent's health comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1. A higher score indicates better health state.
Time Frame: Baseline, Year 1
Population: All enrolled participants who received at least one dose of study drug and had evaluable EQ-5D-5L data. EQ-5D-5L data was not collected during the JADA originating study, zero participants analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JADZ 4 Milligram (mg) Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 450 | 1088 | 171 | 383 | 108 | 305 | 221 | 0
score on a scale
  UK | 0.28 (0.26) | 0.23 (0.24) | 0.19 (0.26) | 0.20 (0.23) | 0.21 (0.22) | 0.19 (0.24) | 0.20 (0.26) |
  US | 0.19 (0.18) | 0.16 (0.17) | 0.13 (0.18) | 0.14 (0.16) | 0.14 (0.15) | 0.13 (0.16) | 0.14 (0.18) |

39. Secondary Outcome: Change From Baseline of Originating Study in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Health State Scores
Description: as for outcome 38
Time Frame: Baseline, Year 3
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 386 | 952 | 146 | 309 | 80 | 219 | 190 | 0
score on a scale
  UK | 0.33 (0.24) | 0.24 (0.25) | 0.20 (0.26) | 0.21 (0.26) | 0.21 (0.22) | 0.22 (0.25) | 0.24 (0.24) |
  US | 0.23 (0.17) | 0.17 (0.17) | 0.15 (0.18) | 0.15 (0.18) | 0.14 (0.15) | 0.15 (0.17) | 0.17 (0.17) |

40. Secondary Outcome: Change From Baseline of Originating Study in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Health State Scores
Description: as for outcome 38
Time Frame: Baseline, Year 5
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 330 | 820 | 122 | 264 | 70 | 169 | 127 | 0
score on a scale
  UK | 0.35 (0.24) | 0.26 (0.26) | 0.19 (0.25) | 0.20 (0.26) | 0.21 (0.22) | 0.22 (0.30) | 0.25 (0.26) |
  US | 0.24 (0.16) | 0.18 (0.18) | 0.13 (0.17) | 0.14 (0.18) | 0.15 (0.15) | 0.15 (0.20) | 0.18 (0.18) |

41. Secondary Outcome: Change From Baseline of Originating Study in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Scores (Self-Perceived Health)
Description: The European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) is a standardized measure of health status of the participant. The second component is a self-perceived health score which is assessed using a VAS that ranged from 0 to 100 millimeter (mm), where 0 mm indicated the worst health you can imagine and 100 mm indicated the best health you can imagine.
Time Frame: Baseline, Year 1
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 450 | 1088 | 171 | 383 | 108 | 305 | 221 | 0
millimeter (mm) | 24.69 (28.50) | 19.72 (28.17) | 15.13 (26.78) | 18.32 (26.35) | 20.96 (24.53) | 14.98 (30.21) | 18.47 (27.31) |

42. Secondary Outcome: Change From Baseline of Originating Study in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Scores (Self-Perceived Health)
Description: as for outcome 41
Time Frame: Baseline, Year 3
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 386 | 952 | 146 | 309 | 80 | 219 | 190 | 0
mm | 28.48 (29.88) | 22.10 (28.02) | 16.29 (25.37) | 16.48 (30.24) | 23.53 (24.70) | 18.79 (30.03) | 21.45 (29.64) |

43. Secondary Outcome: Change From Baseline of Originating Study in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Scores (Self-Perceived Health)
Description: as for outcome 41
Time Frame: Baseline, Year 5
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 330 | 820 | 122 | 264 | 70 | 169 | 127 | 0
mm | 31.13 (28.15) | 23.93 (28.45) | 13.82 (29.59) | 19.34 (27.48) | 26.19 (27.09) | 23.57 (31.67) | 27.31 (27.19) |

44. Secondary Outcome: Percentage of Participants Maintaining a Clinical Disease Activity Index Score (CDAI) ≤10
Description: The CDAI is a tool for measurement of disease activity in RA that does not require a laboratory component and was scored by the investigative site. It integrates TJC28 (scored 0-28 with higher scores indicating higher disease activity), SJC28 (scored 0-28 with higher scores indicating higher disease activity), Patient's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity), and Physician's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity). The CDAI is calculated by summing the values of the 4 components. CDAI scores range from 0 to 76; lower scores indicated lower disease activity. A negative change from baseline indicates improvement in condition.
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 81.6 [77.6 to 85.0] | 75.3 [72.6 to 77.9] | 68.6 [61.3 to 75.2] | 69.9 [65.1 to 74.4] | 52.5 [42.8 to 61.9] | 50.7 [44.8 to 56.6] | 73.3 [67.0 to 78.9] | 60.3 [49.2 to 70.4]

45. Secondary Outcome: Percentage of Participants Maintaining a Clinical Disease Activity Index Score (CDAI) ≤10
Description: as for outcome 44
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 73.3 [68.8 to 77.3] | 67.7 [64.8 to 70.5] | 60.4 [52.8 to 67.4] | 60.4 [55.3 to 65.3] | 49.5 [40.0 to 59.1] | 44.5 [38.8 to 50.4] | 61.4 [54.7 to 67.8] | 56.4 [45.4 to 66.9]

46. Secondary Outcome: Percentage of Participants Maintaining a Clinical Disease Activity Index Score (CDAI) ≤10
Description: as for outcome 44
Time Frame: Years 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 61.6 [56.8 to 66.1] | 61.1 [58.1 to 64.0] | 51.5 [44.0 to 58.9] | 54.6 [49.5 to 59.7] | 44.6 [35.2 to 54.3] | 35.4 [30.0 to 41.2] | 21.9 [16.8 to 28.0] | 56.4 [45.4 to 66.9]

47. Secondary Outcome: Percentage of Participants Maintaining a Clinical Disease Activity Index Score (CDAI) ≤ 2.8
Description: as for outcome 44
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 44.9 [40.2 to 49.7] | 28.3 [25.7 to 31.2] | 21.9 [16.3 to 28.7] | 25.1 [21.0 to 29.8] | 16.8 [10.8 to 25.3] | 13.5 [10.0 to 18.1] | 22.9 [17.7 to 29.0] | 14.1 [8.1 to 23.5]

48. Secondary Outcome: Percentage of Participants Maintaining a Clinical Disease Activity Index Score (CDAI) ≤2.8
Description: as for outcome 44
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 40.1 [35.5 to 44.9] | 30.0 [27.3 to 32.8] | 21.9 [16.3 to 28.7] | 23.5 [19.4 to 28.1] | 22.8 [15.7 to 31.9] | 15.0 [11.2 to 19.7] | 18.6 [13.9 to 24.4] | 20.5 [13.0 to 30.8]

49. Secondary Outcome: Percentage of Participants Maintaining a Clinical Disease Activity Index Score (CDAI) ≤2.8
Description: as for outcome 44
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 33.9 [29.5 to 38.6] | 25.0 [22.5 to 27.8] | 19.5 [14.3 to 26.2] | 22.4 [18.4 to 27.0] | 15.8 [10.0 to 24.2] | 12.8 [9.3 to 17.2] | 8.1 [5.1 to 12.6] | 19.2 [12.0 to 29.3]

50. Secondary Outcome: Percentage of Participants Maintaining a Health Assessment Questionnaire Disability Index (HAQ-DI) Improvement ≥0.22
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate HAQ-DI scores, which ranged from 0 (no disability) to 3 (worst disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition. An improvement of 0.22 or 0.3 points on the HAQ-DI has been identified as a minimal clinically important difference in Rheumatoid Arthritis participants.
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 89.7 [86.5 to 92.3] | 81.4 [78.9 to 83.7] | 78.7 [71.9 to 84.2] | 75.4 [70.7 to 79.5] | 74.3 [65.0 to 81.8] | 69.3 [63.6 to 74.5] | 80.0 [74.1 to 84.8] | 48.7 [37.9 to 59.6]

51. Secondary Outcome: Percentage of Participants Maintaining a Health Assessment Questionnaire Disability Index (HAQ-DI) Improvement ≥0.22
Description: as for outcome 50
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 75.4 [71.1 to 79.3] | 70.4 [67.6 to 73.1] | 64.5 [57.0 to 71.3] | 63.4 [58.3 to 68.2] | 56.4 [46.7 to 65.7] | 54.4 [48.5 to 60.2] | 68.1 [61.5 to 74.0] | 47.4 [36.7 to 58.4]

52. Secondary Outcome: Percentage of Participants Maintaining a Health Assessment Questionnaire Disability Index (HAQ-DI) Improvement ≥0.22
Description: as for outcome 50
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 65.2 [60.5 to 69.6] | 58.5 [55.5 to 61.5] | 51.5 [44.0 to 58.9] | 51.4 [46.3 to 56.4] | 50.5 [40.9 to 60.0] | 39.4 [33.8 to 45.3] | 20.0 [15.2 to 25.9] | 39.7 [29.6 to 50.8]

53. Secondary Outcome: Percentage of Participants Maintaining a Health Assessment Questionnaire Disability Index (HAQ-DI) Improvement ≥0.3
Description: as for outcome 50
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 85.4 [81.7 to 88.5] | 75.6 [72.9 to 78.1] | 72.8 [65.6 to 78.9] | 69.4 [64.5 to 73.9] | 65.3 [55.7 to 73.9] | 61.7 [55.8 to 67.2] | 75.2 [69.0 to 80.6] | 43.6 [33.1 to 54.6]

54. Secondary Outcome: Percentage of Participants Maintaining a Health Assessment Questionnaire Disability Index (HAQ-DI) Improvement ≥0.3
Description: as for outcome 50
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 72.6 [68.1 to 76.6] | 64.8 [61.8 to 67.6] | 61.5 [54.0 to 68.5] | 58.5 [53.4 to 63.4] | 50.5 [40.9 to 60.0] | 47.8 [42.0 to 53.7] | 63.8 [57.1 to 70.0] | 38.5 [28.4 to 49.6]

55. Secondary Outcome: Percentage of Participants Maintaining a Health Assessment Questionnaire Disability Index (HAQ-DI) Improvement ≥0.3
Description: as for outcome 50
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 62.8 [58.0 to 67.3] | 53.4 [50.3 to 56.4] | 46.7 [39.4 to 54.3] | 46.2 [41.1 to 51.3] | 46.5 [37.1 to 56.2] | 35.0 [29.6 to 40.9] | 19.5 [14.7 to 25.4] | 34.6 [25.0 to 45.7]

56. Secondary Outcome: Change From Baseline of Originating Study in Bone Erosion Score
Description: The joint erosion score is a summary of erosion severity in 32 joints of the hands and 12 joints of the feet. The maximum erosion score for a hand joint is 5 and for a foot joint is 10. Thus, the maximal erosion score is 280 for a timepoint (160 for both hands/ wrists and 120 for both feet).
  Each joint is scored according to the surface area involved from 0 to 5 for hand joints and 0 to 10 for the foot joints. The highest score (5 for the hand and 10 for the foot) indicates extensive loss of bone from more than one half of the articulating bone. A score of 0 in either the hand or foot joints indicates no erosion.
  LSM was calculated using an MMRM model with treatment, baseline value, visit, and the interactions of baseline-by-visit and treatment-by-visit as fixed factors.
Time Frame: Baseline, Year 1
Population: as for outcome 32
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

57. Secondary Outcome: Change From Baseline of Originating Study in Bone Erosion Score
Description: as for outcome 56
Time Frame: Baseline, Year 3
Population: as for outcome 33
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 387 | 943 | 137 | 301 | 0 | 0 | 203 | 0
score on a scale | 0.85 [0.63 to 1.08] | 0.92 [0.76 to 1.07] | 0.59 [0.30 to 0.89] | 0.69 [0.49 to 0.89] |  |  | 0.68 [0.32 to 1.03] |

58. Secondary Outcome: Change From Baseline of Originating Study in Bone Erosion Score
Description: as for outcome 56
Time Frame: Baseline, Year 5
Population: as for outcome 34
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 349 | 870 | 127 | 276 | 0 | 0 | 0 | 0
score on a scale | 1.04 [0.77 to 1.32] | 1.18 [0.98 to 1.38] | 0.65 [0.28 to 1.01] | 0.98 [0.74 to 1.23] |  |  |  |

59. Secondary Outcome: Healthcare Resource Utilization
Description: Number of visits to medical care providers related to treatment of Rheumatoid Arthritis (RA) outside of the clinical study. Reported here are healthcare consultations and emergency room consultations from end of originating study to end of participation in study JADY.
Time Frame: Baseline up to 84 Months
Population: All enrolled participants who received at least one dose of study drug and had access to and utilized healthcare services outside of the clinical study.
Measure: Number; unit: consultations
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 451 | 1090 | 180 | 403 | 117 | 331 | 221 | 83
consultations
  Healthcare Consultations | 3134 | 11108 | 2160 | 4573 | 2380 | 5410 | 717 | 749
  Emergency Room Consultations | 95 | 244 | 52 | 131 | 73 | 154 | 40 | 16

60. Secondary Outcome: Percentage of Participants Maintaining a Simplified Disease Activity Index (SDAI) ≤11
Description: SDAI is a tool for measurement of disease activity in RA that integrates TJC28, SJC28, acute phase response using C-reactive protein (milligrams per liter), Patient's Global Assessment of Disease Activity using visual analog scale (cm), and Physician's Global Assessment of Disease Activity using visual analog scale (cm). The SDAI is calculated by summing the values of the 5 components. Lower scores indicated less disease activity.
  The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst). Low disease activity is defined as a SDAI score ≤11.
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 81.6 [77.6 to 85.0] | 75.2 [72.5 to 77.8] | 70.4 [63.1 to 76.8] | 69.1 [64.2 to 73.6] | 53.5 [43.8 to 62.9] | 53.6 [47.7 to 59.5] | 72.4 [66.0 to 78.0] | 59.0 [47.9 to 69.2]

61. Secondary Outcome: Percentage of Participants Maintaining a Simplified Disease Activity Index (SDAI) ≤11
Description: as for outcome 60
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 73.3 [68.8 to 77.3] | 67.8 [64.9 to 70.6] | 60.9 [53.4 to 68.0] | 62.3 [57.2 to 67.1] | 48.5 [39.0 to 58.1] | 44.5 [38.8 to 50.4] | 60.0 [53.3 to 66.4] | 57.7 [46.6 to 68.0]

62. Secondary Outcome: Percentage of Participants Maintaining a Simplified Disease Activity Index (SDAI) ≤11
Description: as for outcome 60
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 61.3 [56.6 to 65.9] | 61.2 [58.2 to 64.1] | 51.5 [44.0 to 58.9] | 53.3 [48.2 to 58.3] | 46.5 [37.1 to 56.2] | 35.4 [30.0 to 41.2] | 23.3 [18.1 to 29.5] | 57.7 [46.6 to 68.0]

63. Secondary Outcome: Percentage of Participants Maintaining a Simplified Disease Activity Index (SDAI) ≤3.3
Description: SDAI is a tool for measurement of disease activity in RA that integrates TJC28, SJC28, acute phase response using C-reactive protein (milligrams per liter), Patient's Global Assessment of Disease Activity using visual analog scale (cm), and Physician's Global Assessment of Disease Activity using visual analog scale (cm). The SDAI is calculated by summing the values of the 5 components. Lower scores indicated less disease activity.
  The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst). Disease remission is defined as an SDAI score of ≤3.3.
Time Frame: Year 1 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 45.3 [40.6 to 50.1] | 28.9 [26.2 to 31.8] | 24.3 [18.4 to 31.2] | 23.5 [19.4 to 28.1] | 13.9 [8.4 to 21.9] | 13.1 [9.6 to 17.7] | 22.9 [17.7 to 29.0] | 14.1 [8.1 to 23.5]

64. Secondary Outcome: Percentage of Participants Maintaining a Simplified Disease Activity Index (SDAI) ≤3.3
Description: as for outcome 63
Time Frame: Year 3 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 39.9 [35.3 to 44.6] | 29.8 [27.1 to 32.6] | 22.5 [16.8 to 29.4] | 21.6 [17.7 to 26.1] | 19.8 [13.2 to 28.6] | 13.5 [10.0 to 18.1] | 15.7 [11.4 to 21.2] | 21.8 [14.1 to 32.2]

65. Secondary Outcome: Percentage of Participants Maintaining a Simplified Disease Activity Index (SDAI) ≤3.3
Description: as for outcome 63
Time Frame: Year 5 after entry into JADY
Population: All enrolled participants who received at least one dose of study drug and completed at least 48 weeks in study JADY.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JADZ 4 mg Baricitinib | JADV 4 mg Baricitinib | JADX 2 mg Baricitinib | JADX 4 mg Baricitinib | JADW 2 mg Baricitinib | JADW 4 mg Baricitinib | JAGS 4 mg Baricitinib | JADA 4 mg Baricitinib
Number analyzed (Participants) | 419 | 1034 | 169 | 366 | 101 | 274 | 210 | 78
percentage of participants | 34.8 [30.4 to 39.5] | 24.7 [22.1 to 27.4] | 20.7 [15.3 to 27.4] | 21.3 [17.4 to 25.8] | 13.9 [8.4 to 21.9] | 11.3 [8.1 to 15.6] | 8.1 [5.1 to 12.6] | 21.8 [14.1 to 32.2]

66. Secondary Outcome: Percentage of Participants With Relapse Event During the 96-Week Step-Down Period
Description: Relapse is defined as a Clinical Disease Activity Index score > 10. The CDAI is a tool for measurement of disease activity in RA that does not require a laboratory component and was scored by the investigative site. It integrates TJC28 (scored 0-28 with higher scores indicating higher disease activity), SJC28 (scored 0-28 with higher scores indicating higher disease activity), Patient's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity), and Physician's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity). The CDAI is calculated by summing the values of the 4 components. CDAI scores range from 0 to 76; lower scores indicated lower disease activity.
  Total number of participants at risk multiplied by estimate of cumulative event probability would need to be rounded up or down to get a whole number.
Time Frame: Week 0 through Week 96 of Step-down
Population: All enrolled participants who were randomized and received at least one dose of study drug during the step-down period for Studies JADX, JADV, JADW, and JAGS.
Measure: Number; unit: percentage of participants
Groups:
- 2 mg Baricitinib Step-down: 2 mg Baricitinib administered orally once daily throughout the 96-week step-down period.
- 4 mg Baricitinib Step-down: 4 mg Baricitinib administered orally once daily throughout the 96-week step-down period.
Arm/Group | 2 mg Baricitinib Step-down | 4 mg Baricitinib Step-down
Number analyzed (Participants) | 498 | 498
percentage of participants
  Week 12 | 11.8 | 5.4
  Week 24 | 26.0 | 12.5
  Week 36 | 31.0 | 18.2
  Week 48 | 36.0 | 21.1
  Week 60 | 41.0 | 26.6
  Week 72 | 45.1 | 29.1
  Week 84 | 46.7 | 31.0
  Week 96 | 47.8 | 34.5

ADVERSE EVENTS:
Time Frame: Baseline up to 84 months
Description: All enrolled participants who received at least 1 dose of study drug and did not discontinue the study for the reason 'Lost to Follow-up' at the first postbaseline visit in study JADY.
  Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- 2 mg Baricitinib: 2 mg Baricitinib administered orally once daily throughout the 84-month treatment period.
- 4 mg Baricitinib: 4 mg Baricitinib administered orally once daily throughout the 84-month treatment period.
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | 2 mg Baricitinib Step-Down | 4 mg Baricitinib Step-Down
All-Cause Mortality (participants affected / at risk) | 7/297 | 70/2579 | 4/592 | 4/594
Serious Adverse Events (participants affected / at risk) | 112/297 | 517/2579 | 164/592 | 178/594
Other Adverse Events (participants affected / at risk) | 234/297 | 1532/2579 | 270/592 | 315/594
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 2 mg Baricitinib (N=297) | 4 mg Baricitinib (N=2579) | 2 mg Baricitinib Step-Down (N=592) | 4 mg Baricitinib Step-Down (N=594)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 2 (2) | 3 (5)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (5) | 7 (7) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 5 (5) | 1 (1) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 11 (13) | 1 (1) | 3 (4)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (3) | 1 (1) | 1 (1) | 2 (5)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 4 (4) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 3 (6) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 4 (6) | 2 (3) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Congenital central nervous system anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0/66 (0) | 1/548 (1) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Adrenal suppression (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 6 (13) | 3 (4) | 1 (1)
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal perforation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Macular rupture (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 6 (7) | 1 (1) | 0 (0)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol interaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 4 (5) | 3 (3) | 3 (5)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 8 (9) | 1 (1) | 10 (10)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 4 (4)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone tuberculosis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 5 (6) | 2 (3) | 5 (7)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bursitis infective staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 12 (14) | 0 (0) | 4 (5)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Cytomegalovirus hepatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3) | 4 (4) | 3 (3) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Extrapulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fascial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 7 (7) | 1 (1) | 2 (2)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
H1n1 influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 5 (5) | 15 (20) | 2 (3) | 5 (5)
Herpes zoster infection neurological (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Histoplasmosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Infective aneurysm (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Meningoencephalitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0/66 (0) | 1/548 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Paracoccidioides infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Plasmodium falciparum infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasmodium vivax infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 15 (17) | 34 (36) | 10 (14) | 12 (15)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia cryptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 1 (2)
Pneumonia legionella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 2 (5) | 2 (2) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Salpingitis (Infections and infestations) | 0/231 (0) | 1/2031 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (4) | 10 (10) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular abscess (Infections and infestations) | 0 (0) | 0 (0) | 1/152 (1) | 0/146 (0)
Thrombophlebitis septic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (7) | 12 (12) | 0 (0) | 3 (4)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 4 (6) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vulvitis (Infections and infestations) | 0 (0) | 0 (0) | 1/440 (2) | 0/448 (0)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Crush injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epiphyseal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 13 (14) | 1 (1) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 7 (8) | 3 (3) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 1 (1) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (2) | 3 (3) | 2 (3) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Keratorhexis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0) | 1 (3)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 7 (7) | 0 (0) | 1 (1)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Open globe injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 6 (6) | 1 (1) | 1 (1)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (5) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1) | 4 (7)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram t wave inversion (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza a virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mycobacterium tuberculosis complex test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (8) | 1 (3) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (5) | 3 (6) | 6 (7)
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7) | 5 (7) | 2 (2)
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (5) | 1 (2) | 1 (1)
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (13) | 42 (56) | 6 (9) | 5 (5)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 (6) | 16 (18) | 0 (0) | 3 (3)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (2) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaplastic meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/231 (0) | 1/2031 (1) | 1/440 (2) | 0/448 (0)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/231 (0) | 1/2031 (1) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0) | 1 (2)
Extranodal marginal zone b-cell lymphoma (malt type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Giant cell tumour of tendon sheath (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Large intestine fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (4) | 2 (2) | 0 (0)
Lung adenocarcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mueller's mixed tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/231 (0) | 1/2031 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nonkeratinising carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/231 (0) | 1/2031 (1) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/231 (1) | 2/2031 (2) | 0/440 (0) | 1/448 (2)
Ovarian cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/231 (0) | 1/2031 (1) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/231 (1) | 0/2031 (0) | 0 (0) | 0 (0)
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/66 (2) | 3/548 (3) | 2/152 (2) | 0/146 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0/152 (0) | 1/146 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0/152 (0) | 1/146 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/231 (0) | 1/2031 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the parotid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1/440 (1) | 0/448 (0)
Uterine carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1/440 (1) | 0/448 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/231 (0) | 2/2031 (3) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Central nervous system vasculitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fistula (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 5 (7) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 9 (10) | 1 (1) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/231 (1) | 2/2031 (2) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/231 (0) | 1/2031 (1) | 1/440 (1) | 0/448 (0)
Device dislocation (Product Issues) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Device failure (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device loosening (Product Issues) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 3 (5) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (3) | 4 (4) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Iga nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 5 (5) | 3 (3) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 6 (7) | 0 (0) | 1 (3)
Urinary tract inflammation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adnexa uteri cyst (Reproductive system and breast disorders) | 0/231 (0) | 2/2031 (2) | 0 (0) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0/440 (0) | 1/448 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/66 (0) | 1/548 (1) | 0 (0) | 0 (0)
Cervical cyst (Reproductive system and breast disorders) | 0/231 (0) | 1/2031 (2) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2/440 (2) | 1/448 (2)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0/440 (0) | 1/448 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0/231 (0) | 1/2031 (1) | 0 (0) | 0 (0)
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0/440 (0) | 1/448 (1)
Endometriosis (Reproductive system and breast disorders) | 0/231 (0) | 1/2031 (1) | 2/440 (2) | 0/448 (0)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0/231 (0) | 4/2031 (5) | 0/440 (0) | 1/448 (3)
Ovarian cyst (Reproductive system and breast disorders) | 0/231 (0) | 3/2031 (4) | 0/440 (0) | 1/448 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0/152 (0) | 1/146 (1)
Uterine polyp (Reproductive system and breast disorders) | 0/231 (0) | 1/2031 (1) | 0/440 (0) | 1/448 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1/231 (1) | 0/2031 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/231 (1) | 0/2031 (0) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0/231 (0) | 1/2031 (2) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 9 (17) | 2 (11) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6) | 1 (1) | 2 (3)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 18 (21) | 5 (5) | 3 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Respite care (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Finger amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1/440 (1) | 0/448 (0)
Internal fixation of fracture (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Limb reconstructive surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scar excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal cyst excision (Surgical and medical procedures) | 0/231 (0) | 1/2031 (1) | 0 (0) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 14 (16) | 2 (3) | 4 (4)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (5) | 3 (3) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Necrosis ischaemic (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosed varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg Baricitinib (N=297) | 4 mg Baricitinib (N=2579) | 2 mg Baricitinib Step-Down (N=592) | 4 mg Baricitinib Step-Down (N=594)
Anaemia (Blood and lymphatic system disorders) | 18 (21) | 126 (156) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 20 (24) | 72 (79) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 18 (25) | 87 (107) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 16 (17) | 56 (62) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 48 (65) | 291 (431) | 44 (61) | 65 (91)
Herpes zoster (Infections and infestations) | 30 (32) | 160 (167) | 39 (42) | 53 (57)
Influenza (Infections and infestations) | 15 (16) | 147 (176) | 30 (35) | 56 (64)
Nasopharyngitis (Infections and infestations) | 42 (95) | 291 (488) | 54 (109) | 58 (101)
Pharyngitis (Infections and infestations) | 19 (30) | 119 (181) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 17 (19) | 66 (71) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 23 (31) | 100 (121) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 58 (106) | 281 (454) | 46 (54) | 51 (63)
Urinary tract infection (Infections and infestations) | 53 (84) | 241 (336) | 34 (48) | 52 (72)
Blood creatine phosphokinase increased (Investigations) | 22 (26) | 176 (229) | 20 (26) | 33 (44)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 16 (19) | 142 (162) | 18 (18) | 32 (32)
Hyperlipidaemia (Metabolism and nutrition disorders) | 18 (20) | 133 (157) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 (58) | 155 (229) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 42 (55) | 162 (181) | 35 (41) | 36 (43)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (25) | 53 (63) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 27 (38) | 141 (250) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 19 (21) | 90 (106) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 16 (16) | 47 (50) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (46) | 105 (134) | 35 (37) | 25 (32)
Hypertension (Vascular disorders) | 33 (36) | 196 (218) | 38 (38) | 46 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT01885078/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT01885078/SAP_001.pdf